CLINICAL TRIAL: NCT02503787
Title: A Prospective, Multi-center, Open-label Study of Programming Options in Spinal Cord Stimulation.
Brief Title: OPTIONS Spinal Cord Stimulation Programming Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1675
Record Dates: First submitted 2015-07-14; First posted 2015-07-21 (Estimated); Results first posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-08

CONDITIONS: Pain, Intractable
Keywords: chronic pain; intractable pain; failed back surgery syndrome
MeSH Terms: conditions — Pain, Intractable; Chronic Pain; Failed Back Surgery Syndrome | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label treatment (Other): Spinal Cord Stimulation (SCS)
  Interventions: Device: Spinal Cord Stimulation (SCS)

INTERVENTIONS:
Device: Spinal Cord Stimulation (SCS) — SCS programming options

SUMMARY:
The purpose of this study is to evaluate programming options in spinal cord stimulation for the management of chronic, intractable pain of the trunk and limbs.

DETAILED DESCRIPTION:
Prospective, multi-center, open-label study evaluating programming options in spinal cord stimulation on pain relief. All eligible subjects will undergo a Spinal Cord Stimulation (SCS) device trial that includes an intraoperative programming trial. Subjects experiencing a positive response to the programming parameters (improvement in average overall pain relief) during the trial from baseline will move forward with a permanent implant. Those not reporting a positive response to the programming parameters will be exited from the study.

The subjects will complete a number of assessment worksheets to characterize their Quality of Life and function and the level of pain they are experiencing from the baseline to 3 months post neurostimulation trial.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for Spinal Cord Stimulation (SCS) system (trial and implant) per labeled indication(back and leg pain)
* Willing and able to provide a signed and dated informed consent
* At least 18 years old at the time of informed consent
* Willing and able to attend visits and comply with the study protocol
* Capable of using the patient programmer and recharging the neurostimulator
* Willing to not increase pain medications from baseline through the 3-Month Visit

Exclusion Criteria:

* Currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound study results.
* Psychological or other health conditions that would interfere with the subject's ability to fulfill the requirements of the protocol.
* Trialed or implanted with SCS, subcutaneous stimulation, peripheral nerve stimulation or an implantable intrathecal drug delivery system
* Implanted with a cardiac device (e.g., pacemaker, defibrillator)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: OPTIONS Clinical Research Study Team, Study Director — Medtronic Implantable Therapies
Locations (11):
- United States (11):
  - Valley Pain Consultants-North Scottsdale, Scottsdale, Arizona
  - Synovation Medical Group, Chula Vista, California
  - Center for Interventional Pain Spine, Wilmington, Delaware
  - Pain Care LLC, Stockbridge, Georgia
  - Millennium Pain Center, Bloomington, Illinois
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - St. Luke's Neurosurgical Associates, Bethlehem, Pennsylvania
  - Precision Spine Care, Tyler, Texas
  - Swedish Pain Services, Seattle, Washington
  - Northwest Pain Care, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled subjects will undergo a Spinal Cord Stimulation device trial that includes an intraoperative programming trial. Subjects experiencing a positive response (improvement in average overall pain relief) during the trial will move forward with a permanent implant. Those not reporting a positive response will be exited from the study.
Period: Enrollment
Arm/Group | Open Label Treatment
Started | 64
Completed | 44
Not Completed | 20
Not completed — Withdrawal by Subject | 6
Not completed — Inclusion/exclusion criteria not met | 4
Not completed — Physician Decision | 2
Not completed — Insurance issue | 2
Not completed — Lost to Follow-up | 1
Not completed — Study closure | 1
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Inability to implant system | 1
Not completed — Unable to be programmed | 1
Period: Device Trial (HD Programming Trial)
Arm/Group | Open Label Treatment
Started | 44
Completed | 37
Not Completed | 7
Not completed — Lack of Efficacy | 6
Not completed — Withdrawal by Subject | 1
Period: Successful Trial (≥50% Pain Relief)
Arm/Group | Open Label Treatment
Started | 37
Completed | 32
Not Completed | 5
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 2
Period: Implant to 3 Month Endpoint
Arm/Group | Open Label Treatment
Started | 32
Completed | 29
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Implanted and Device Activated subjects
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32
Average Overall Pain [Mean (Standard Deviation); unit: units on a scale] — Self reported daily average overall pain score 5 days prior to baseline. The question is scored 0-10 (0=no pain; 10=pain as bad as can be).
  units on a scale | 7.5 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Overall Pain as Measured by the Diary-reported Numeric Pain Rating Scale (NPRS) Questionnaire
Description: Self reported daily average overall pain score 5 days prior to baseline and at 3 months post device activation in subjects receiving programming options in spinal cord stimulation. The question is scored 0-10 (0=no pain; 10=pain as bad as can be).
Time Frame: From baseline to 3 months post device activation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 32
units on a scale | -3.7 (2.3)
Statistical Analysis 1: Comparison: Open Label Treatment; A negative value for change in pain represents a reduction (improvement) of the subject's pain score. The null hypothesis was that the mean change from baseline to 3 months equals 0. The sample provided over 90% power, with two-sided significance level of 0.05, to detect a change of 2 points; Test type: Superiority; p < 0.01, t-test, 2 sided

2. Secondary Outcome: Patient Global Impression of Change
Description: Evaluate study subject impression of change as measured by the Patient Global Impression of Change questionnaire. The questionnaire encompasses change in ACTIVITY LIMITATIONS, SYMPTOMS, EMOTIONS, and OVERALL QUALITY OF LIFE, scored on a scale of 1-7 (1=no change or the condition has gotten worse: 7=A great deal better, and a considerable improvement that has made all the difference).
Time Frame: From baseline to 3 months post device activation
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 32
Participants
  7 - A great deal better | 10
  6 - Better | 12
  5 - Moderately better | 6
  4 - Somewhat better | 1
  3 - A little better | 1
  2 - Almost the same | 2
  1 - No change (or worse) | 0

3. Other Pre Specified Outcome: Change in Average Back Pain as Measured by the Diary-reported Numeric Pain Rating Scale (NPRS) Questionnaire
Description: Self reported daily average back pain score 5 days prior to baseline and at 3 months post device activation in subjects receiving programming options in spinal cord stimulation. The question is scored 0-10 (0=no pain; 10=pain as bad as can be).
Time Frame: From baseline to 3 months post device activation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 32
units on a scale | -3.8 (2.0)

4. Other Pre Specified Outcome: Change in Average Leg Pain as Measured by the Diary-reported Numeric Pain Rating Scale (NPRS) Questionnaire
Description: Self reported daily average leg pain score 5 days prior to baseline and at 3 months post device activation in subjects receiving programming options in spinal cord stimulation. The question is scored 0-10 (0=no pain; 10=pain as bad as can be).
Time Frame: From baseline to 3 months post device activation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 32
units on a scale | -4.1 (2.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning at the device trialing procedure and throughout implant and the 3 month activation phase.
Description: The sample for adverse event reporting is the 48 subjects who initiated the device trialing procedure (44 subjects started the HD programming trial). Device, therapy, and/or procedure-related adverse events were collected. Adverse events that were documented as the reason for discontinuation were also collected regardless of etiology.
Groups:
- Device: Neurostimulator: RestoreSensor SureScan MRI Rechargeable Neurostimulator
  RestoreSensor SureScan MRI Rechargeable Neurostimulator: RestoreSensor SureScan MRI Rechargeable Neurostimulator
Arm/Group | Device: Neurostimulator
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 1/48
Other Adverse Events (participants affected / at risk) | 12/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device: Neurostimulator (N=48)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) — Pain in Bilateral Feet
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device: Neurostimulator (N=48)
Paraesthesia (uncomfortable sensation) (Nervous system disorders) | 7 (9)
Implant site warmth (General disorders) | 5 (5)
Pain (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restrictions on the PI allow for the sponsor to review results communications prior to public release and to embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to sponsor for review. The sponsor is also allowed to require changes for technical correctness and to protect confidential information, copyrightable or patentable material; and when reasonably requested, extend the embargo up to an additional 90 days.